CLINICAL TRIAL: NCT03547778
Title: Efficacy of Vaginal Misoprostol For Pain Relief During Office Hysteroscopy and Endometrial Biopsy; A Double Blind Randomized Controlled Trial
Brief Title: Misoprostol in Office Hysteroscopy and Endometrial Biopsy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to get patients interested in the study
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00034137
Record Dates: First submitted 2018-05-22; First posted 2018-06-06 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2019-03

CONDITIONS: Office Hysteroscopy and Endometrial Biopsy
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Intervention Model Description: A Double Blind Randomized Controlled Trial
Who Masked: Participant, Care Provider
Masking Description: The participants and the care providers (performing the procedure) will not know about the randomization. The research coordinator will perform the randomization and the medicine dispensed by the pharmacy. The study drug and placebo are similar looking, hence the participants and providers would not be able to identify them.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Misoprostol group (Experimental): Patients in this arm will receive vaginal misoprostol (50 mcg), the night before the procedure (concurrent office hsyteroscopy and endometrial biopsy).
  Interventions: Drug: Misoprostol 50 mcg pesssary
- Placebo group (Placebo Comparator): Participants in this group will receive placebo (fatty acid), which looks similar to misoprostol and has to be inserted vaginally the night before the procedure.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Misoprostol 50 mcg pesssary — Participants in the study arm will receive vaginal misoprostol (50 mcg) to be inserted the night before the procedure. Whereas the control group will get a placebo.
  Arms: Misoprostol group
Drug: Placebos — The control group will receive placebo pessaries to be inserted vaginally the night before the procedure.
  Arms: Placebo group

SUMMARY:
We hypothesize that use of vaginal misoprostol will help in reducing the pain scores when used prior to concurrent office hysteroscopy and endometrial biopsy in a particular subgroup of women who are anticipated to require cervical dilatation.

DETAILED DESCRIPTION:
Office hysteroscopy (OH) and endometrial biopsy (EMB) is increasingly performed for evaluation of various gynecologic conditions. It has replaced traditional dilatation and curettage for evaluation of intrauterine pathology. It is more acceptable to most women as it is quick, safe and cost effective with higher diagnostic accuracy. However, pain encountered at the time of procedure is a major limitation and at times lead to incomplete procedure. The variables that influence women's experience of pain during these procedures are nulliparity, menopausal status, pre-existing anxious state, use of tenaculum, presence of synechiae in the cervical canal, and duration of procedure.

The average pain score recorded at the end of procedures when OH and EMB were performed simultaneously was 7 on a 10 cm VAS scale (Visual analogue scale) 5 among pre and post menopausal women who received pre-procedure analgesia in the form of oral Non-Steroidal Anti Inflammatory drug (NSAID) and application of local anesthetic gel. Among patients where only intracervical topical anesthetic injection was used, the pain score at the end of OH and EMB was 9.22 (low pain) and 11.52 (moderate pain), respectively, on a 20cm VAS. Most women describe EMB as "moderately" or "severely" painful6. A significant source of pain during endometrial sampling is placement of tenaculum on the cervix. Interventions that have been studied to reduce pain with EMB include misoprostol for cervical ripening, intrauterine lidocaine infusion, paracervical block, and pre-procedure NSAIDs. The results are variable with modest benefit on pain with only an intrauterine lidocaine infusion with or without NSAID or/and misoprostol. Similarly, during OH also, there are multiple points where women experience pain. It can be during tenaculum placement, introduction of the hysteroscope, distension of uterine cavity, intrauterine procedures, and withdrawal of scope. Out of many interventions evaluated, local anesthesia via paracervical block provided consistent decreases in intraoperative and postoperative pain scores. There were mixed data on efficacy of intracervical blocks and no evidence to support the use of intrauterine anesthesia or topical gels, sprays, or creams. Premedication with opioid analgesics or NSAIDs do not confer benefit in pain management during office hysteroscopy. Misoprostol for cervical ripening prior to diagnostic hysteroscopy neither reduce pain nor facilitate the procedure for hysteroscopes with diameters of less than 6 mm in premenopausal women, but there may be a benefit in postmenopausal women. In contrast, another systematic review examining use of misoprostol before hysteroscopy found that misoprostol given to premenopausal women reduced the need for cervical dilatation and the incidence of cervical laceration.

Misoprostol is a prostaglandin E1 analog that was first marketed in the 1980s to prevent gastric ulcer. It can be administered sublingually, orally, vaginally, or rectally. Peak serum levels are achieved after vaginal administration. The plasma concentration increases gradually after vaginal administration, reaching its maximum level after 70-80 minutes. Misoprostol is commonly used in gynecology for inducing dilatation of the cervix for termination of pregnancy and removing retained products of conception. It helps in non-pregnant women to dilate the cervix and provides easy access to the uterine cavity for transcervical procedures such as hysteroscopy and intrauterine device placement. To evaluate the optimal dose of vaginal misoprostol for cervical priming before operative hysteroscopy, low dose (200mcg) and high dose (400 mcg) misoprostol was compared in a recent randomized control trial. They found no difference in perioperative dilatation time, and subjective difficulty of cervical dilatation assessed by surgeons. However, the incidence of misoprostol related adverse events such as abdominal pain, pre-insertion nausea and cramping were less in the group who received 200 mcg misoprostol. But it is important to note that even 200 mcg misoprostol is associated with 50% incidence of abdominal cramping. Since we would be conducting outpatient diagnostic procedures only, we propose that use of 50 mcg misoprostol would lead to adequate cervical dilatation to successfully complete the OH and EMB with lower incidence of associated complications (abdominal cramping, vaginal bleeding, and nausea). Moreover, it is important to note that the standard operating procedure of the fibroid and endometriosis center has been the administration of 50 mcg misoprostol to patients undergoing simultaneous OH and EMB. This practice that has been ongoing for over 12 months has provided very favorable results. No other study has evaluated the efficacy of such a low dose and it would be interesting to explore the minimal effective dose, which can be used for simultaneous OH and EMB to yield effective results in terms of lower pain scores and lower incidence of associated complications. As mentioned previously, studies evaluating the role of misoprostol in alleviating overall pain during OH and EMB had mixed reviews. But those studies have been performed in the general population. It is important to note that there are subgroups of women (previous cesarean section, nulliparous, postmenopausal, previous loop surgery) who more often need dilatation of the cervix to facilitate passage of the hysteroscope. Therefore, this trial will focus on these subgroups to assess whether the use of prostaglandin analogue provides clinically significant reduction in pain, reduces the need for dilatation and incidence of genital trauma and whether these benefits outweigh the potential harms (bleeding, laceration, abdominal cramping, fever etc.)

ELIGIBILITY:
Inclusion Criteria:

All consecutive female patients aged 18-70 years presenting to the Center for successive OH and EMB with the ability to provide written informed consent and meets at least one of the criteria mentioned below:

* Previous cesarean section
* Nulliparous
* Postmenopausal
* Previous loop electrosurgical excision procedure (LEEP) or cone biopsy
* Previous myomectomy

Exclusion Criteria:

Premenopausal multiparous women with no prior surgeries performed on the uterus.

* Patients unable to provide informed consent
* Patients visiting the fibroid and endometriosis center with abnormal uterine bleeding, infertility or for preoperative evaluation; however, OH and EMB is not required for their evaluation based on their providers' clinical judgment.
* Patients with genital tract lesions.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Pain score recorded in VAS | Day of procedure
  The current study aims to evaluate if vaginal misoprostol (50 mcg) administered prior to Office hysteroscopy and endometrial biopsy when performed successively in the same office visit decreases overall pain perception during the procedure among subgroup of women who are anticipated to have difficult entry into the cervical canal

SECONDARY OUTCOMES:
Cervical dilatation | Day of procedure
  We intend to investigate whether vaginal misoprostol use reduces the need for dilatation and eventually helps in successfully completing the procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Department of Obstetrics and Gynecology, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cicinelli E, Didonna T, Ambrosi G, Schonauer LM, Fiore G, Matteo MG. Topical anaesthesia for diagnostic hysteroscopy and endometrial biopsy in postmenopausal women: a randomised placebo-controlled double-blind study. Br J Obstet Gynaecol. 1997 Mar;104(3):316-9. doi: 10.1111/j.1471-0528.1997.tb11460.x. PMID 9091008
- [Background] Urman RD, Punwani N, Bombaugh M, Shapiro FE. Safety considerations for office-based obstetric and gynecologic procedures. Rev Obstet Gynecol. 2013;6(1):e8-e14. PMID 23687556